CLINICAL TRIAL: NCT05550155
Title: Efficacy of Maintenance Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment in Reducing Auditory Verbal Hallucinations (AVH) With High Frequency and Neuronavigation Guidance: A Double-blind, Randomized and Multicentric Study
Brief Title: Efficacy of Maintenance Repetitive Transcranial Magnetic Stimulation (rTMS) in Auditory Verbal Hallucinations
Acronym: MAINSTIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 21-0157
Record Dates: First submitted 2022-09-19; First posted 2022-09-22 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Schizophrenia; Psychosis
Keywords: Transcranial Magnetic Stimulation; Auditory verbal Hallucination; Neuronavigation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations | interventions — Transcranial Magnetic Stimulation; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sham rTMS (Sham Comparator): The sham treatment, following the group assignment, will be maintained during the two successive phases of the evaluated protocol. One initial sham rTMS phase will consist of four sham stimulation sessions (20 Hz sham) within two consecutive days. One sham rTMS maintenance phase will consist of two sham stimulation sessions on one day every week for one month and then every two weeks for three months.
  Clinical data will be assessed by an investigator blind to group assignment until the end of the study. Patients will also be blind to stimulation. A questionnaire will assess the investigator physician and patient beliefs about what group the patient was involved in (placebo group or active group) at the end of the treatment initial phase and at the end of the treatment maintenance phase
  Interventions: Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS)
- active rTMS (Experimental): The active treatment, following the group assignment, will be maintained during the two successive phases of the evaluated protocol. One initial active rTMS phase will consist of four stimulation sessions (20 Hz) within two consecutive days. One active rTMS maintenance phase will consist of two active stimulation sessions on one day every week for one month and then every two weeks for three months.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation (rTMS) Treatment — a 4-month maintenance procedure of active rTMS
  Arms: active rTMS
Device: Sham Repetitive Transcranial Magnetic Stimulation (rTMS) — a 4-month maintenance procedure of sham rTMS
  Arms: sham rTMS

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) can alleviate persistent auditory verbal hallucinations (AVH) in schizophrenic patients, but the classical procedure with low-frequency stimulation for several weeks upon the left temporoparietal junction have shown modest therapeutic effects, and there is currently no robust predictive factor to the response of the treatment. In a previous multicentric, randomized, and double-blind controlled study, it has been demonstrated that a high-frequency rTMS over an anatomical target can rapidly affect AVHs. Moreover, an intensification of the classical procedure delivering 20-Hz rTMS over a 2-day period was used in addition to a personalized anatomical stimulation target and neuronavigation guidance. Besides the significant efficacy of the procedure, the efficacy was maximal at two weeks after the end of the treatment. In this project, the hypothesis is that the two-day cure could benefit from maintenance rTMS sessions every week for one month and then every two weeks for 3 months to provide an optimal strategy for a long-lasting AVH reduction. This has for now never been tested. Predictive factors to the response of the treatment are also investigated.

DETAILED DESCRIPTION:
To investigate the clinical efficacy of a 4-month maintenance procedure of rTMS in AVH reduction, a multicenter, controlled, double-blind study enrolling 120 patients randomly assigned in two groups is proposed. The active group will receive active rTMS with a two-day intense procedure (consisting in 4 20-Hz rTMS sessions within two days) and a maintenance phase with a two- rTMS session every week for one month and then every two weeks the next 3 months (i.e. 24 rTMS sessions). The individual target will be personalized and guided by neuronavigation. The placebo group will benefit from the exact same procedure but with sham rTMS instead of active rTMS. Patients will be carried out during 5 months and what distinguishes responders from non-responders will be studied. Among other variables, BDNF serum levels as a reflect of the individual neural plasticity and the measurement of the scalp-to-cortex distance to the target as a reflect of the cerebral morphological interindividual variations will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female; Age ≥ 18 years ≤ 65 years
* Diagnosis of schizophrenia or schizoaffective disorders according to DSM 5.0 criteria
* Patients treated with at least one antipsychotic medication
* Presence of auditory verbal hallucinations despite the optimization of the antipsychotic dosage for at least 6 weeks. This will be operationalized by a minimum AHRS score > 10
* Stable medication dosage for at least 6 weeks before the rTMS treatment
* Patient who understands the French language
* The agreement of the curatorship or tutorship in the case of a protected adult
* Willing to comply with scheduled visits, as outlined in the protocol
* Covered by, or having the right to Social Security or European cover
* Informed and written consent

Exclusion Criteria:

* Women who are pregnant
* Patients with contraindications for rTMS (history of epilepsy, neurologic stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid derivation, metallic splinters in the eyes)
* Patients included or planning to be included in another medical research protocol
* Patients unable to complete the protocol follow-up
* Any brain pathological abnormality known or diagnosed by the cerebral MRI
* Contre-indication for cerebral MRI (metallic fix tooth prosthesis, neurologic stimulator, pacemaker, cardiac defibrillator, cardiac prosthesis, vascular prosthesis, intracranial clips or clamps, cerebrospinal fluid derivation, metallic splinters in the eyes, severe claustrophobia)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-10-30 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
the number of times a patient is assessed as a responder | between baseline and month 5
  the number of times a patient is assessed as a responder in the active versus the sham group during their follow-up between baseline (D1) and at the end of the maintenance treatment (M5), i.e. the month after the last maintenance session.

CONTACTS AND LOCATIONS:
Overall Officials: Sonia Dollfus, Principal Investigator — University Caen Normandie
Locations (1):
- Caen University Hospital, Caen, France